CLINICAL TRIAL: NCT04051385
Title: Assesment of Gingival Crevicular Fluid and Serum ErbB4/Neuregulin-4 Levels in Periodontal Disease and Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Sadiye Gunpinar, Asst. Prof., Abant Izzet Baysal University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017/113; 2018.06.05.1310 (Other Grant/Funding Number: Bolu Abant Izzet Baysal University Research Foundation)
Record Dates: First submitted 2019-08-07; First posted 2019-08-09 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Periodontitis
Keywords: periodontal disease; gingival crevicular fluid; macrophage; ErbB-4; neuregulin-4
MeSH Terms: conditions — Periodontitis; Periodontal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- stage II grade B periodontitis (Active Comparator): GCF and serum samples were taken before and after treatment from stage II grade B periodontitis patients.
  Intervention: Non- surgical periodontal treatment (SRP and oral hygiene instructions)
  Interventions: Other: non surgical periodontal treatment; Other: Gingival crevicular fluid and serum collection
- stage III grade B periodontitis (Active Comparator): GCF and serum samples were taken before and after treatment from stage III grade B periodontitis patients.
  Intervention: Non- surgical periodontal treatment (SRP and oral hygiene instructions)
  Interventions: Other: non surgical periodontal treatment; Other: Gingival crevicular fluid and serum collection
- gingivitis (Active Comparator): GCF and serum samples were taken before and after treatment from gingivitis patients.
  Intervention: Non- surgical periodontal treatment (Scaling and oral hygiene instructions)
  Interventions: Other: non surgical periodontal treatment; Other: Gingival crevicular fluid and serum collection
- periodontally healthy (Placebo Comparator): GCF and serum samples were taken at baseline from periodontally healthy individuals.
  Interventions: Other: Gingival crevicular fluid and serum collection

INTERVENTIONS:
Other: non surgical periodontal treatment — SRP under local anaesthesia, in a total of 2 clinical visits. Oral hygiene instructions including the modified Bass technique and an appropriate interdental cleaning device with dental floss and interdental brush.
  Arms: gingivitis; stage II grade B periodontitis; stage III grade B periodontitis
Other: Gingival crevicular fluid and serum collection — GCF with filter paper using the intracrevicular method and serum collection

SUMMARY:
This study aimed to investigate gingival crevicular fluid (GCF) and serum ErbB4 and Nrg4 levels in periodontal health and disease. A total of 80 individuals, 20 patients with stage II grade B periodontitis, 20 patients with stage III grade B periodontitis, 20 with gingivitis and 20 periodontally healthy individuals were included. Whole-mouth and site-specific clinical periodontal parameters including probing depth, clinical attachment level, bleeding on probing, gingival index, plaque index and papillar bleeding index were recorded. GCF and serum ErbB4 and Nrg4 levels were measured by enzyme-linked immunosorbent assay. Statistical analysis was performed by using non-parametric tests.

DETAILED DESCRIPTION:
A total of 80 individuals, comprising 20 patients with stage II grade B periodontitis (P1 Group), 20 patients with stage III grade B periodontitis (P2 Group), 20 patients with gingivitis (G Group), and 20 periodontally healthy controls (H Group) were involved in the study.

The participants were classified into four groups depending on periodontal health status in accordance with the consensus reports of the 2017 World Workshop:

1. periodontally healthy (H) group: no interproximal attachment loss (AL), probing depth (PD) ≤3 mm, bleeding on probing (BOP) scores <10%;
2. gingivitis (G) group: no interproximal AL, PD ≤3 mm, and BOP ≥10%;
3. stage II grade B periodontitis (P1) group: 3 <PD ≤5 mm and 3 ≤ clinical attachment loss (CAL) <5 mm in one or more sites of the 2 non-adjacent teeth in at least two quadrants of the mouth, full mouth BOP ≥ 10% and no tooth loss due to periodontitis
4. stage III grade B periodontitis (P2) group: PD >5 mm and CAL ≥ 5 mm in one or more sites of the 2 non-adjacent teeth in at least two quadrants of the mouth, full mouth BOP >10% and tooth loss due to periodontitis of ≤4 teeth.

Inclusion criteria were as follows:

1. aged >18 years,
2. having at least 16 natural teeth (excluding third molar),
3. not having any diagnosed medical illness or drug intake that could affect the periodontal condition.

Exclusion criteria were as follows:

1. The patients who had taken antibiotics, nonsteroidal antiinflammatory or any other drugs within the past 3 months,
2. received nonsurgical or surgical periodontal treatment,
3. a restorative and endodontic therapy requirement,
4. a removable partial denture and/or having orthodontic therapy
5. Current pregnancy or lactation, obesity, heavy smoking and having serum C reactive protein (CRP) > 3mg/L.

All individuals were examined at baseline and four weeks after non-surgical periodontal treatment including, whole mouth probing depth (PD), CAL, presence of bleeding on probing (BOP), papillar bleeding index (PBI), gingival index (GI) and plaque index (PI) except the third molars. PD and CAL were measured at six sites per tooth using a manual periodontal probe.

The non-surgical periodontal treatment for P1 and P2 groups included supra- and subgingival scaling, root planing and oral hygiene instructions. Subgingival scaling and root planing were performed under local anesthesia in two sessions within the 48-72 h. Gingivitis group had supra-and subgingival scaling, polishing and oral hygiene instructions. The treatment of gingivitis and periodontitis patients were performed by a periodontist (BM) using hand and ultrasonic instruments. All measurements were performed by the same calibrated examiner (BM).

Gingival crevicular fluid (GCF) sampling

GCF samples were obtained from four nonadjacent interproximal sites in two maxillar and two mandibular multi-rooted teeth by standardized filter paper strips. GCF samples were taken from four sites with GI <1, PD ≤ 3, PBI =0 and CAL =0 in the H group; from four sites with GI ≥2, PD ≤3, PBI >2 and CAL=0 in the G group; from four sites (deepest pockets 3 <PD ≤5) with GI ≥2, PBI >2 and 3 ≤CAL <5 mm in P1 group; and from four sites (deepest pockets PD ≥5) with GI ≥2, PBI >2 and CAL ≥5 mm in P2 group according to the baseline clinical measurements.

Serum sampling

Serum samples were taken following GCF sampling before the periodontal treatment. Six milliliters of venous blood were obtained by a standard venipuncture method and the serum was separated from blood by centrifugation at 1,500 g for 20 minutes.

Biochemical Assays

Levels of GCF ErbB4, Nrg4, IL-6, IL-10 and levels of serum ErbB4, Nrg4, nitric oxide synthase (NOS)2 and Arg1 were measured by the enzyme-linked immunosorbent assay (ELISA) using commercial kits according to the manufacturer's guidelines.

Statistical Analysis

All data analyses were performed using a statistical software package. Comparisons of clinical and biochemical parameters between the study groups were performed using the Kruskal- Wallis with Mann Whitney U test with Bonferroni correction method. The intragroup comparisons (at baseline and first month) were performed using Wilcoxon test for paired samples. Associations among levels of the GCF and serum biomarkers and clinical parameters were also examined using the Spearman rank correlation analysis.

ELIGIBILITY:
Inclusion Criteria:

* Aged >18 years,
* Having at least 16 natural teeth (excluding third molar),
* Not having any diagnosed medical illness or drug intake that could affect the periodontal condition.

Exclusion Criteria:

* Patients who had taken antibiotics, nonsteroidal antiinflammatory or any other drugs within the past 3 months,
* Patients received nonsurgical or surgical periodontal treatment,
* Patients who have a restorative and endodontic therapy requirement,
* Having a removable partial denture and/or having orthodontic therapy,
* Current pregnancy or lactation,
* Obesity,
* Heavy smoking and having serum CRP > 3mg/L .

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2019-01-18 (Actual); Study Completion 2019-01-18 (Actual)

PRIMARY OUTCOMES:
Biochemical parameters (ErbB4 and Nrg4) | Baseline and 4 weeks after treatment
  The changes in levels of ErbB4 and Nrg4, four weeks after periodontal treatment determined by ELISA.
  The changes in levels of ErbB4 and Nrg4 were analyzed to determine as a diagnostic biomarker of periodontal disease.
Biochemical parameters (IL-6, IL-10, nitric oxide synthase (NOS) 2 and Arg1) | Baseline and 4 weeks after treatment
  The changes in GCF levels of IL-6 and IL-10 and serum levels of nitric oxide synthase (NOS)2 and Arg1, four weeks after periodontal treatment determined by ELISA.

SECONDARY OUTCOMES:
Probing pocket depth | Baseline and 4 weeks after treatment
  The changes in probing pocket depth was measured for determining of the severity of disease and clinical outcome
Clinical attachment loss | Baseline and 4 weeks after treatment
  The changes in clinical attachment loss was measured for determining the severity of disease
Gingival index | Baseline and 4 weeks after treatment
  Gingival index was recorded for classifying and evaluating sulcular gingival inflammation. Gingival index was also analyzed to detect the relationship between ErbB4/Nrg4 and periodontal disease.
Plaque index | Baseline and 4 weeks after treatment
  Plaque index was recorded for determining and classifying oral hygiene status
Bleeding on probing | Baseline and 4 weeks after treatment
  Bleeding on probing was recorded for classifying and evaluating gingival inflammation especially for apically sulcular inflammation. This was also analyzed to detect the relationship between ErbB4/Nrg4 and periodontal disease.
Papillar bleeding index | Baseline and 4 weeks after treatment
  Papillar bleeding index was recorded for classifying and evaluating the papillar gingival inflammation. This index was also analyzed to detect the relationship between ErbB4/Nrg4 and periodontal disease.

CONTACTS AND LOCATIONS:
Overall Officials: Sadiye Gunpinar, Asst. Prof., Principal Investigator — Abant Izzet Baysal University
Locations (1):
- Bolu Abant Izzet Baysal University, Bolu, Turkey (Türkiye)

REFERENCES:
- [Background] Papapanou PN, Sanz M, Buduneli N, Dietrich T, Feres M, Fine DH, Flemmig TF, Garcia R, Giannobile WV, Graziani F, Greenwell H, Herrera D, Kao RT, Kebschull M, Kinane DF, Kirkwood KL, Kocher T, Kornman KS, Kumar PS, Loos BG, Machtei E, Meng H, Mombelli A, Needleman I, Offenbacher S, Seymour GJ, Teles R, Tonetti MS. Periodontitis: Consensus report of workgroup 2 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. J Periodontol. 2018 Jun;89 Suppl 1:S173-S182. doi: 10.1002/JPER.17-0721. PMID 29926951
- [Background] Caton JG, Armitage G, Berglundh T, Chapple ILC, Jepsen S, Kornman KS, Mealey BL, Papapanou PN, Sanz M, Tonetti MS. A new classification scheme for periodontal and peri-implant diseases and conditions - Introduction and key changes from the 1999 classification. J Clin Periodontol. 2018 Jun;45 Suppl 20:S1-S8. doi: 10.1111/jcpe.12935. PMID 29926489